CLINICAL TRIAL: NCT07098247
Title: Exploring Photon-Counting CT for Enhanced Target Delineation and Dose Accuracy in Personalized Radiotherapy - ANTHEM
Acronym: RAD4/RT_ANTHEM
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: RAD4/RT_ANTHEM
Record Dates: First submitted 2025-04-22; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patient with cancer: 500 patients undergoing radiotherapy for orphan cancers, chronic conditions, and anatomically complex regions such as brain, head and neck, thorax, liver, pancreas and pelvis.

SUMMARY:
Radiotherapy remains a cornerstone of oncology care, particularly for rare or orphan cancers and chronic oncologic and rare non oncologic conditions, where precision and individualized treatment planning are necessary. Advances in imaging technologies are crucial to overcome the challenges posed by these cases, especially in achieving accurate tumor delineation and dose delivery. Photon-counting CT (PCCT) represents a transformative step forward in imaging technology. Unlike conventional energy-integrating CT, PCCT offers a) superior spatial resolution, enabling clearer visualization of tumor margins and fine anatomical structures, b) enhanced tissue characterization, allowing better differentiation between tumor tissues and normal tissue; c) spectral imaging capabilities, facilitating improved dose calculations. These attributes are particularly advantageous in high-precision radiotherapy techniques, such as stereotactic body radiotherapy (SBRT) or proton therapy, where small errors in target delineation or dose delivery can significantly impact treatment outcomes. However, very limited data reporting the clinical use of PCCT for RT planning are available.

ELIGIBILITY:
Inclusion criteria:

* ≥18 years old patients
* tumors located in challenging anatomical regions (brain, head and neck, liver, pancreas prostate), or Cardiac disease requiring RT by photon or proton at our Institution.

Exclusion criteria:

- 18 years old patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing radiotherapy for orphan cancers, chronic conditions, and anatomically complex regions such as brain, head and neck, thorax, liver, pancreas and pelvis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Improve RT target delineation accuracy and differentiation of organs-at-risk (OARs). | day 1 (day of simulation TC)
  During the simulation, the investigator will evaluate the image quality obtained from photon-counting TC imaging compared to conventional imaging techniques, and assess how this improved imaging could enhance radiotherapy treatment planning. The data will be evaluated by indicative scores of imaging quality and treatement planning.
  minimum scale value is one and indicates a poor quality of the imaging - maximum scale value is five and indicates excellent image quality

SECONDARY OUTCOMES:
Enhanced dose calculation precision, particularly for proton therapy | Day 1 (day of simulation TC)
  During the simulation, the investigator will evaluate the image quality obtained from photon-counting TC imaging compared to conventional imaging techniques, and assess how this improved imaging could enhance radiotherapy treatment planning. The data will be evaluated by indicative scores of imaging quality and treatement planning.
  minimum scale value is one and indicates a poor quality of the imaging - maximum scale value is five and indicates excellent image quality

CONTACTS AND LOCATIONS:
Overall Officials: Marta Scorsettti, MD, radiation oncologist, Principal Investigator — Humanitas University
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, Milan, Italy